CLINICAL TRIAL: NCT01093846
Title: A 38-week Extension to a 24 Week Multicenter, Randomized, Double-masked, Placebo Controlled Study to Assess the Difference in the Rate of Recurrent Exacerbations in Behçet's Patients With Posterior or Panuveitis Treated With AIN457 vs Placebo Adjunctive to Standard-of-care Immunosuppressive Therapy (SHIELD Study)
Brief Title: 38 Week Extension Study to CAIN457C2303
Acronym: SHIELD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Core Study in Behcet's disease with mostly active uveitis did not meet its primary endpoint
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457C2303E1; 2009-013901-33
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Uveitis
Keywords: uveitis
MeSH Terms: conditions — Uveitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- AIN457 300 mg every 2 weeks (Experimental)
  Interventions: Drug: AIN457
- AIN457 300 mg monthly (Experimental)
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo AIN457

INTERVENTIONS:
Drug: AIN457 — 300mg every 4 weeks
  Arms: AIN457 300 mg monthly
Drug: AIN457 — 300mg every 2 weeks
  Arms: AIN457 300 mg every 2 weeks
Drug: Placebo AIN457 — Placebo to AIN457
  Arms: Placebo

SUMMARY:
A 38-week extension to a 24 week multicenter, randomized, double-masked, placebo controlled study to assess the difference in the rate of recurrent exacerbations in Behçet's patients with posterior or panuveitis treated with AIN457 vs placebo adjunctive to standard-of-care immunosuppressive therapy

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Novartis Investigative Site, Baltimore, Maryland, United States
- Novartis Investigative Site, Alexandria, Egypt
- Novartis Investigative Site, Grenoble, France
- Novartis Investigative Site, Heidelberg, Germany
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Lin-Ko, Taiwan
- Novartis Investigative Site, Sfax, Tunisia
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Altindag / Ankara
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 300 mg Every 2 Weeks: 300 mg every two weeks
- AIN457 300 mg Monthly: 300 mg monthly
Period: Overall Study
Arm/Group | AIN457 300 mg Every 2 Weeks | AIN457 300 mg Monthly | AIN457 Placebo
Started | 19 | 18 | 22
Completed | 0 | 0 | 1
Not Completed | 19 | 18 | 21
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4
Not completed — Condition no longer required study drug | 1 | 1 | 1
Not completed — Administrative Problems | 18 | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 300 mg Every 2 Weeks | AIN457 300 mg Monthly | AIN457 Placebo | Total
Number analyzed (Participants) | 19 | 18 | 22 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (10.01) | 36.8 (13.07) | 34.9 (11.20) | 36.0 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11 | 22
  Male | 13 | 13 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Continuous Treatment With Subcutaneous AIN457 Compared to Placebo in Reducing the Rate of Recurrent Ocular Exacerbations in Behçet's Patients With Intermediate Uveitis, Posterior Uveitis or Panuveitis in Group 1.
Description: The primary objective of the study was to determine the effect of continuous treatment with subcutaneous AIN457 compared to placebo in reducing the rate of recurrent ocular exacerbations in Behçet's patients with intermediate uveitis, posterior uveitis or panuveitis in patients who completed the core study and continued treatment in the extension study (Group 1).Due to early termination of the study AIN457C2303E1, the analysis of extension period was changed. No efficacy analyses were completed, the safety analyses are available in the summary of AEs which occurred during the extension and safety follow-up periods and are shown in the safety section .
Time Frame: 62 weeks
Arm/Group | Early Termination
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- AIN457 300mg Every 2 Weeks: AIN457 300mg every 2 weeks. Safety is provided over the entire treatment period. This includes the core and extension period.
- AIN457 300mg Monthly: AIN457 300mg monthly Safety is provided over the entire treatment period. This includes the core and extension period.
- Placebo: Placebo Safety is provided over the entire treatment period. This includes the core and extension period.
Arm/Group | AIN457 300mg Every 2 Weeks | AIN457 300mg Monthly | Placebo
Serious Adverse Events (participants affected / at risk) | 7/39 | 8/39 | 5/39
Other Adverse Events (participants affected / at risk) | 28/39 | 27/39 | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=39) | AIN457 300mg Monthly (N=39) | Placebo (N=39)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract cortical (Fellow eye) (Eye disorders) | 0 | 0 | 1
Cataract nuclear (Fellow eye) (Eye disorders) | 0 | 0 | 1
Cataract subcapsular (Fellow eye) (Eye disorders) | 0 | 0 | 1
Choroiditis (Fellow eye) (Eye disorders) | 1 | 0 | 0
Glaucoma (Fellow eye) (Eye disorders) | 0 | 0 | 1
Retinal infiltrates (Fellow eye) (Eye disorders) | 1 | 0 | 0
Retinal infiltrates (Study eye) (Eye disorders) | 1 | 0 | 0
Uveitis (Fellow eye) (Eye disorders) | 1 | 1 | 0
Uveitis (Study eye) (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Behcet's syndrome (Immune system disorders) | 0 | 1 | 0
Behcet's syndrome (Fellow eye) (Immune system disorders) | 0 | 1 | 0
Behcet's syndrome (Study eye) (Immune system disorders) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0
Hypopyon (Fellow eye) (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intraocular pressure increased (Fellow eye) (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=39) | AIN457 300mg Monthly (N=39) | Placebo (N=39)
Cataract subcapsular (Fellow eye) (Eye disorders) | 4 | 1 | 0
Cataract subcapsular (Study eye) (Eye disorders) | 4 | 1 | 1
Eye pain (Study eye) (Eye disorders) | 1 | 2 | 2
Retinal vasculitis (Study eye) (Eye disorders) | 2 | 0 | 1
Vision blurred (Fellow eye) (Eye disorders) | 0 | 6 | 1
Vision blurred (Study eye) (Eye disorders) | 0 | 2 | 3
Visual acuity reduced (Study eye) (Eye disorders) | 4 | 2 | 1
Vitreous floaters (Study eye) (Eye disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 2
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 3
Fatigue (General disorders) | 2 | 2 | 4
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Oedema peripheral (General disorders) | 3 | 2 | 0
Pyrexia (General disorders) | 6 | 3 | 4
Conjunctivitis infective (Study eye) (Infections and infestations) | 1 | 2 | 1
Influenza (Infections and infestations) | 2 | 4 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Rash pustular (Infections and infestations) | 2 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Blood glucose increased (Investigations) | 0 | 2 | 0
Intraocular pressure increased (Study eye) (Investigations) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 9 | 7 | 10
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study AIN457C2303E1, the analysis of extension period was changed. No efficacy analyses were completed, the safety analyses were reduced to summary of AEs occurred during the extension and safety follow-up periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.